CLINICAL TRIAL: NCT04640129
Title: A Multicentre Clinical Trial in HBsAg Seroclearance After Receiving Combined Therapy of Peginterferon and Tenofovir in Nucleos(t)Ide Analogue-treated Patients With HBV Related Liver Fibrosis.
Brief Title: HBsAg Seroclearance in Adults With HBV Related Liver Fibrosis After Receiving Combined Therapy of Peg-IFN and Tenofovir.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL15
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDF group (Active Comparator): tenofovir 300mg taken orally per day.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- peg-IFN-α plus TDF group (Experimental): peg-IFN-α 180ug given subcutaneous injection per week combined with tenofovir 300mg taken orally per day .
  Interventions: Drug: PEG-Interferon Alfa, Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: PEG-Interferon Alfa, Tenofovir Disoproxil Fumarate — Combination therapy group was treated with PEG-interferon Alfa in addition to TDF monotherapy
  Arms: peg-IFN-α plus TDF group
Drug: Tenofovir Disoproxil Fumarate — TDF monotherapy
  Arms: TDF group

SUMMARY:
Liver fibrosis caused by hepatitis B virus (HBV) infection is easy to progress to liver cirrhosis and liver cancer, with great harm and poor therapeutic effect. Nucleos(t)ide analogues (NAs) are the most commonly anti-HBV drugs currently . Long-term use of NAs can inhibit HBV DNA and achieve the purpose of reducing poor prognosis. However, adverse prognosis, such as liver cirrhosis and liver cancer, cannot be completely eliminated even under the status of virologic inhibition under THE action of NAs. Current studies have shown that the lower the HBV surface antigen (HBsAg) is, the better the long-term prognosis is. As another anti-HBV drug, pegylated-interferon-α (peg-IFN-α) has the immune regulation effect that NAs do not have, which can bring irreplaceable effects in HBsAg reduction and liver fibrosis reversal. Therefore, the combined therapy of NAs and peg-IFN-α is a hot issue in the field of liver diseases over the world, but the research and application of the combined therapy in patients with liver fibrosis are very few. The preliminary results of our previous research showed that the combined therapy of peg-IFN-α and NAs in patients with HBV related fibrosis were safe, and had a significant effect on HBsAg decline. On this basis, this study intends to carry out a multicentre, non-randomized concurrent controlled trial, comparing the safety and efficacy between combined therapy (peg-IFN-α plus tenofovir) and tenofovir monotherapy in patients with liver fibrosis, especially focusing on HBsAg's decline and clearance, and the improvement of liver fibrosis degree, in order to find a better therapy, and to guide the clinical decision making.

ELIGIBILITY:
Inclusion Criteria:

* 1.Positive hepatitis b surface antigen; 2.Infection of hepatitis b virus DNA > 0.5 year before anti-HBV treatment; 3.Receiving treatment of nucleoside/nucleotide analogues at least one year before recruited; 4.Age from 18 to 55 years old; 5.Normal liver function(ALT<ULN,AST<ULN and TBil<ULN); 6.Undetectable hepatitis b virus DNA or less than 100IU/ml; 7.Liver biopsy suggested fibrosis of liver into F1~F3(Metavir score system) or LSM between 6 and 12 kpa measured by fibroscan; 8.Liver ultrasound: normal or echo thickening, and portal vein diameter ≤ 12mm.

Exclusion Criteria:

* 1.Decompensated cirrhosis, hepatocellular carcinoma or other malignancy; 2.Pregnancy, lactation or female has plan of pregnancy within 18 months; 3.Accompanied with other active liver diseases(HAV, HCV, HDV, HEV, autoimmune liver disease, drug-induced liver injury, alcoholic liver disease, genetic metabolic liver disease, etc.)； 4.Accompanied with human immunodeficiency virus infection or congenital immune deficiency diseases; 5.Accompanied with severe diabetes, autoimmune diseases etc. and other important organ dysfunctions; 6.Patients who fail to comply with this research arrangement and sign an informed consent form; 7.Patients can not follow-up; 8.Investigator considering inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 336 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
proportion of HBsAg seroclearance/seroconversion | 48 weeks
  proportion of seroclearance or seroconversion of HBV surface antigen compared with baseline

SECONDARY OUTCOMES:
proportion of HBsAg seroclearance/seroconversion | 96 weeks
  Proportion of seroclearance or seroconversion of HBV surface antigen compared with baseline
proportion of fibrosis improvement | 96 weeks
  Proportion of patients with improved fibrosis compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu S, Wu L, Mei Y, Liu Z, Lin L, Yuan J, Li J, Li X, Peng L. Prospective, multicentre, randomised controlled trial comparing the seroclearance of HBsAg between combination therapy of peg-interferon alpha and tenofovir with tenofovir monotherapy in nucleos(t)ide analogue-experienced patients with HBV-related liver fibrosis: a study protocol. BMJ Open. 2021 Oct 25;11(10):e049104. doi: 10.1136/bmjopen-2021-049104. PMID 34697111